CLINICAL TRIAL: NCT04254380
Title: An Open-label, Randomized, Multicenter, Phase 3 Study to Compare the Immunogenicity, Efficacy, and Safety of Gan & Lee Insulin Lispro Injection to Humalog in Adult Subjects With Type 1 Diabetes Mellitus (T1DM)
Brief Title: Gan & Lee Evaluation of New Biosimilar for Type 1 Lispro
Acronym: GENTL 1
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: GanLee cancelled study -FDA Draft Guidance: "Clinical Immunogenicity Considerations for Biosimilar & Interchangeable Insulin Products" released 11/25/2019
Sponsor: Gan and Lee Pharmaceuticals, USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GL-LSPT1-3003
Record Dates: First submitted 2020-01-13; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes; Diabetes Type 1; Type 1; Basal; Insulin; Lispro; T1DM; Diabetes Mellitus; Insulin Dependent Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance | interventions — gallium nitrate; Insulin Lispro

STUDY DESIGN:
Intervention Model Description: Subjects who meet the eligibility criteria will be centrally randomized 1:1 in an open-label fashion to receive either Gan & Lee Insulin Lispro Injection or Humalog for 26 weeks. Randomization will be stratified by country.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Gan & Lee Insulin Lispro Injection (Experimental): Gan & Lee Insulin Lispro Injection for subcutaneous injection, 100 U/mL, in a disposable multidose pen injector with a pre-filled 3-mL type I glass cartridge. Subjects randomized to the Gan & Lee Insulin Lispro Injection group will participate in the study for 26 weeks.
  Interventions: Biological: Gan & Lee Insulin Lispro Injection
- Active Comparator: Humalog (Active Comparator): EU-authorized Humalog KwikPen® - insulin lispro injection, solution for subcutaneous injection, 100 U/mL (pre-filled). Subjects randomized to the Humalog group will participate in the study for 26 weeks.
  Interventions: Biological: Humalog

INTERVENTIONS:
Biological: Gan & Lee Insulin Lispro Injection — Route of administration: subcutaneous injection
  Arms: Experimental: Gan & Lee Insulin Lispro Injection
Biological: Humalog — Route of administration: subcutaneous injection
  Arms: Active Comparator: Humalog

SUMMARY:
Primary Objective:

• To compare the immunogenicity of Gan & Lee Insulin Lispro Injection and EU-authorized Humalog following treatment in adult subjects with T1DM

Secondary Objectives:

* To evaluate the safety of Gan & Lee Insulin Lispro Injection in comparison with that of EU authorized Humalog following treatment in adult subjects with T1DM
* To evaluate the efficacy of Gan & Lee Insulin Lispro Injection in comparison with that of EU authorized Humalog following treatment in adult subjects with T1DM

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant, non-lactating female subjects between the ages of 18 and 75 years, inclusive.
2. Female subjects of child-bearing potential, willing to use contraceptive method(s), agreed by the Investigator, to prevent pregnancy during the study.
3. Ability to provide written, personally signed, and dated informed consent to participate in the study, in accordance with the ICH GCP Guideline E6 and all applicable regulations, before initiating any study related procedures.
4. Ability to understand and fully comply with all study procedures and restrictions.
5. A confirmed diagnosis of T1DM and who have been on an approved basal-bolus insulin regimen for at least 6 months prior to Screening. The type or brand of insulins should not have changed in the 6 months before Screening.
6. Do not expect to change the brand or type of their basal insulin during the study.
7. C-peptide ≤ 1.0 ng/mL
8. HbA1c ≤ 10.0%
9. Body mass index (BMI) ≥ 19 kg/m2 and ≤ 35 kg/m2
10. Adherence to a prudent diet and exercise regimen recommended by the medical provider in accordance with local standard of care or American Diabetes Association recommendations, and willingness to maintain this regimen consistently for the duration of the study.

Exclusion Criteria:

1. Participation in another clinical study within 30 days or 5 half-lives of last dose of experimental medication before Screening, whichever is longer.
2. Previous use of Gan & Lee Insulin Lispro Injection.
3. Use of insulin neutral protamine hagedorn or insulin detemir within 6 months prior to study entry.
4. Current or expected use of an insulin pump or use of continuous glucose measurement to monitor blood glucose during the study.
5. Diabetic ketoacidosis (DKA) within 6 months before Screening.
6. Brittle T1DM within 1 year before Screening, defined as more than 2 hospitalizations related to diabetes mellitus (excluding hospitalizations for diagnostic purposes), and/or severe hypoglycemia for which the subject experiences severe cognitive impairment requiring external assistance for recovery.
7. Renal replacement therapy required or with an estimated (or measured) glomerular filtration rate < 15 mL/min (Modification of Diet in Renal Disease calculation).
8. Any clinically significant cardiovascular (CV) or cerebrovascular event, e.g., myocardial infarction (MI), acute coronary syndrome (ACS), recent revascularization (including coronary artery bypass graft procedures [CABG], percutaneous coronary intervention [PCI]), transient ischemic attack (TIA), or hemorrhagic or ischemic stroke within 3 months before Screening.
9. History of congestive heart failure defined as New York Heart Association (NYHA) Stage III or IV.
10. Inadequately controlled or unstable hypertension as defined by a systolic blood pressure (SBP) > 160 mmHg or diastolic blood pressure (DBP) > 100 mmHg at Screening and/or Randomization.
11. Inadequately controlled thyroid disease, as reflected by abnormal TSH and free T4 values. (Hypothyroid or hyperthyroid conditions should be resolved or stabilized before Screening according to local standard of care).
12. Any clinically significant (in the opinion of the Investigator) hematology, chemistry, or urinalysis test results at Screening, including any liver function test > 3X of the upper limit of normal (ULN) or bilirubin > 1.5X of the ULN (subjects with elevated bilirubin due to Gilbert syndrome are eligible to participate, if such tests were performed in the past).
13. Autonomic neuropathy resulting in a diagnosis of gastroparesis.
14. Hemoglobin < 12 g/dL for males or < 11 g/dL for females at Screening.
15. Hospitalization within the 14 days before Screening, or planned hospitalization at any time during the study.
16. Newly prescribed or high-dose (60 mg/day prednisone or equivalent) treatment with glucocorticosteroids, immunosuppressants, or cytostatic agents due to disorders of the immunological system, such as rheumatoid arthritis, psoriasis, spondyloarthritis, and asthma, within 60 days before Screening (Medications under following scenario are allowed: chronically administered oral, inhaled, topical, or intra-articular corticosteroids at a stable dosage; stable therapy with disease modifying agents [e.g., methotrexate, sulfasalazine]; disease is inactive [e.g., remission, well controlled stable phase]; and no significant changes in treatment scheme are expected).
17. History of human immunodeficiency virus (HIV) or Hepatitis B or Hepatitis C infections.
18. Any unresolved infection or a history of active infection within 30 days before screening other than mild viral illness (as judged by the Investigator).
19. Current use of other medications for diabetes treatment, such as dipeptidyl peptidase 4 inhibitors (DPP4i), glucagon-like peptide 1 receptor agonists (GLP1-R), or sodium glucose cotransporter 2 inhibitors (SGLT2i) (See Appendix 1 [Section 16.1] for a list of prohibited medications).
20. A history of alcohol use of more than two drinks a day on average for the last year, or a history of alcohol or substance abuse within 2 years before Screening.
21. Previous (within 3 months before Screening) or anticipated treatment with interferons.
22. History of malignancy (except for treated non-melanoma skin cancer and treated cervical adenocarcinoma in situ) within 5 years before Screening
23. Receiving blood transfusion or undergoing plasmapheresis within 6 months before Screening.
24. History of splenectomy.
25. Intolerance or history of hypersensitivity to insulin lispro or any excipient of the study drugs.
26. Any other clinically significant medical or psychiatric condition, or one requiring further evaluation that in the opinion of the Investigator could interfere with conduct of the study or interpretation of the data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Treatment developed AIAs or important increase in AIA titers | Week 1 to Week 26
  The percentage of subjects in each treatment group who develop treatment induced AIAs, defined as newly confirmed positive AIA development or important (at least a 4-fold) increase in titers after baseline and up to visit Week 26.

SECONDARY OUTCOMES:
Percentage of subjects with negative AIA at baseline who develop positive AIA after baseline | Week 1 to Week 26
  The percentage of subjects in each treatment group with negative AIA at baseline who develop confirmed positive AIA after baseline and up to visit Week 26.
Percentage of subjects with important increase in titers | Week 1 to Week 26
  The percentage of subjects in each treatment group with confirmed positive AIA at baseline and at least a 4-fold increase in titers after baseline and up to visit Week 26.
Mean change from baseline in AIA titers | Week 1 to Week 26
  The mean change from baseline in each treatment group in AIA titers after baseline and up to visit Week 26.
Percentage of subjects with confirmed positive AIA who develop anti-insulin NAbs | Week 1 to Week 26
  The percentage of subjects in each treatment group with confirmed positive AIA after baseline and up to visit Week 26 who develop any anti-insulin NAbs after baseline and up to visit Week 26.
Percentage of subjects with positive AIA after baseline | Week 1 to Week 26
  The percentage of subjects in each treatment group with confirmed positive AIA after baseline and up to visit Week 26.
Incidence and severity of all treatment-emergent adverse events | Week 1 to Week 26
  The incidence and severity of all treatment-emergent adverse events and the following subgroups:
  Adverse events of special interest. Serious adverse events, including fatal events. Adverse events leading to termination of the study treatment and/or early withdrawal from the study.
  Treatment-related adverse events. IP device-related adverse events. Injection site reactions. The incidence of clinically significant laboratory abnormalities. The incidence of clinically significant abnormalities in physical examination and vital signs.
Change from baseline in HbA1c at visit Week 26 | Week 1 to Week 26
  Change from baseline in HbA1c at visit Week 26 in each treatment group.
Percentage of subjects who achieve an HbA1c of ≤ 7.0% at visit Week 26 | Week 1 to Week 26
  The number and percentage of subjects who achieve an HbA1c of ≤ 7.0% at visit Week 26 in each treatment group.

CONTACTS AND LOCATIONS:
Overall Officials: Jia Lu, PhD, Study Director — Gan & Lee Pharmaceuticals, USA
Locations (107):
- United States (58):
  - Advanced Research Center, Anaheim, California
  - Valley Research, Fresno, California
  - Angel City Research, Inc., Los Angeles, California
  - California Medical Research Association, Northridge, California
  - Mills-Peninsula Health Services, San Mateo, California
  - Care Access Research - Santa Clarita, Santa Clarita, California
  - Metabolic Institute of America, Tarzana, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - IMMUNOe International Research Centers - Longmont, Longmont, Colorado
  - Chase Medical Research of Greater New Haven, Hamden, Connecticut
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - M & O Clinical Research, Fort Lauderdale, Florida
  - Sweet Hope Research Specialty Inc., Hialeah, Florida
  - Homestead Associates in Research, Homestead, Florida
  - Med Research of Florida, Miami, Florida
  - Suncoast Clinical Research - Pasco County, New Port Richey, Florida
  - Florida Institute for Clinical Research, LLC, Orlando, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - Suncoast Clinical Research - Pinellas County, Palm Harbor, Florida
  - Meridien Research - Spring Hill, Spring Hill, Florida
  - Metabolic Research Institute, West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - IACT Health - Columbus Regional Medical Group Endocrine Consultants - Columbus, Columbus, Georgia
  - IACT Health - Columbus Regional Medical Group Endocrine Consultants, Newnan, Georgia
  - Endocrine Research Solutions, Roswell, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Midwest CRC, Crystal Lake, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Kentucky Diabetes Endocrinology Center, Lexington, Kentucky
  - Bay West Endocrinology Associates, Baltimore, Maryland
  - BTC Network - Capital Diabetes and Endocrine Associates - Camp Springs, Camp Springs, Maryland
  - Endocrine & Metabolic Consultants, Rockville, Maryland
  - Quality Clinical Research, Omaha, Nebraska
  - Palm Research Center, Las Vegas, Nevada
  - BTC Network - Garden State Endocrinology - Brick, Brick, New Jersey
  - The Endocrine Group, LLP, Albany, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - University Physicians Group, Staten Island, New York
  - PharmQuest, Greensboro, North Carolina
  - Physicians East - Greenville, Greenville, North Carolina
  - Carteret Medical Group - Morehead City, Morehead City, North Carolina
  - Endocrinology Research Associates, Columbus, Ohio
  - Your Diabetes Endocrine Nutrition Group, Inc., Mentor, Ohio
  - Intend Research, Norman, Oklahoma
  - Lynn Institute of Stillwater, Stillwater, Oklahoma
  - Care Access Research - Warwick, Warwick, Rhode Island
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - Amarillo Medical Specialists, Amarillo, Texas
  - Austin Regional Clinic, Austin, Texas
  - Texas Diabetes & Endocrinology - Central Austin, Austin, Texas
  - Research Institute of Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - El Paso Medical Research Institute, El Paso, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Austin Regional Clinic - Kelly Lane, Pflugerville, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Northeast Clinical Research of San Antonio, Schertz, Texas
  - Crossroads Clinical Research, Victoria, Texas
- Czechia (5):
  - Diabetologie České Budějovice s.r.o, České Budějovice, Jihočeský kraj
  - Diahaza s.r.o., Holešov
  - StefaMed, Hradec Králové
  - Clintrial, Prague
  - Milan Kvapil s.r.o, Prague
- Germany (5):
  - Diabeteszentrum DO, Dortmund
  - Diabetes Schwerpunktpraxis, Duisburg
  - Diabetes-falkensee.de - Zentrum für klinische Studien, Falkensee
  - RED-Institut GmbH, Oldenburg
  - Diabetologische Praxis, Saarlouis
- Hungary (11):
  - Lausmed Egeszsegugyi es Szolgaltato Kft., Baja
  - Dél-pesti Centrumkórház - Országos Hematológiai és Infektológiai Intézet, Budapest
  - Bajcsy-Zsilinszky Kórház és Rendelőintézet, Budapest
  - Trantor 99 Bt Anyagcsere Centrum, Budapest
  - Debreceni Egyetem Kenézy Gyula Egyetemi Kórház, Debrecen
  - Békés Megyei Központi Kórház Pándy Kálmán Tagkórház, Gyula
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Kanizsai Dorottya Kórház, Nagykanizsa
  - Markusovszky Egyetemi Oktatokorhaz, Szombathely
  - Medical-Expert Kutatási - Kísérleti és Szolgáltató Kft, Veszprém
  - Zala Megyei Szent Rafael Kórház, Zalaegerszeg
- Poland (16):
  - Centrum Badań Klinicznych PI-House, Gdansk
  - Niepubliczny Zaklad Opieki Zdrowotnej Gdanska Poradnia Cukrzycowa, Gdansk
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Centrum Medyczne Pratia Katowice, Katowice
  - Pratia MCM Kraków, Krakow
  - NZOZ Medyczne Centrum Diabetologiczno-Endokrynologiczno-Metaboliczne "Diab-Endo-Met", Krakow
  - CenterMed Lublin Sp. z o.o, Lublin
  - KO-MED Centra Kliniczne Lublin - Królewska, Lublin
  - Bogdan Walko Niepubliczny Zakład Opieki Zdrowotnej Przychodnia Specjalistyczna MEDICA, Lublin
  - Centrum Medyczne Grunwald, Poznan
  - Nasz Lekarz Przychodnie Medyczne, Torun
  - AMED Centrum Medyczne, Warsaw
  - Centralny Szpital Kliniczny Ministerstwa Spraw Wewnętrznych i Administracji w Warszawie, Warsaw
  - Centrum Medyczne K2J2, Wołomin
  - Regionalna Poradnia Diabetologiczna, Wroclaw
  - Centrum Medyczne Oporów, Wroclaw
- Spain (12):
  - Complejo Hospitalario Universitario La Coruña (Gerencia de Gestión Integrada de A Coruña), A Coruña
  - Hospital de la Santa Creu i de Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebrón, Barcelona
  - Complejo Hospitalario Universitario de Ferrol, Ferrol
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Ramón Y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Fundació Hospital de l'Esperit Sant, Santa Coloma de Gramenet
  - Nuevas Tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen de Valme, Seville

IPD SHARING:
Plan to Share IPD: No